CLINICAL TRIAL: NCT02542904
Title: Extensive Mesenteric Excision (EME) Versus Local Mesenteric Excision (LME) for Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, Jinling Hospital, Jinling Hospital, China
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: EME vs. LME
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Postoperative Disease Recurrence; Crohns Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- LME (Active Comparator): the anastomosis was performed as stapled side-to-side with local excision of the mesenteric tissue adjacent to the diseased bowel
  Interventions: Procedure: mesenteric excision
- EME (Active Comparator): the anastomosis was performed as a stapled side-to-side anastomosis with extensive excision of mesenteric tissue.
  Interventions: Procedure: mesenteric excision

INTERVENTIONS:
Procedure: mesenteric excision

SUMMARY:
Crohn's patients receiving ileocolonic resection are randomized into extensive mesenteric resection group and local mesenteric resection group.

DETAILED DESCRIPTION:
Randomization was performed intraoperatively once the surgeon had determined that there were no other sites of disease and that either type of anastomosis could be performed safely. Computer generated randomization was carried out within strata using randomized permuted blocks to ensure balance of the groups.

All surgery was performed by a single group of surgeons experienced in the surgical treatment of Crohn's disease. Surgery was performed open or laparoscopically depending on patient factors and surgeon preference. The resection was performed grossly normal resection margins, with side-to-side anastomosis. The presence of mesenteric marginal thickening with confirmation by naked eye assessment of the mucosal aspect of the bowel were used to establish the limits of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease limited to the distal ileum and/or right colon

Exclusion Criteria:

* Concomitant anastomosis/strictureplasty at another site of the gastrointestinal tract, and required a temporary fecal diversion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-08; Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
postoperative endoscopic recurrence | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China